CLINICAL TRIAL: NCT00589602
Title: Phase II Feasibility Study of T-Cell Depletion in Allogeneic Unrelated Bone Marrow Transplantation (MUD ALLO BMT) Followed by Delayed T-Cell Infusions
Brief Title: T-Cell Depletion, Donor Hematopoietic Stem Cell Transplant (HSCT), and T-Cell Infusions in Treating Patients With Hematologic Cancer or Other Diseases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jaroslaw Maciejewski, Department Chair of Translational Hematology and Oncology Research, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCF-6501; P30CA043703 (NIH)
Record Dates: First submitted 2008-01-01; First posted 2008-01-09 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Malignant Plasma Cell Neoplasms; Myelodysplastic Syndromes; Precancerous/Nonmalignant Condition; Secondary Myelofibrosis
Keywords: Adult leukemia; lymphoma; myelodysplastic syndromes; plasma cell disorders
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Myelodysplastic Syndromes; Precancerous Conditions | interventions — Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Intervention Model Description: Allogeneic Hematopoietic Stem Cell Transplantation
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- T-Cell Depletion Transplant (Experimental): Our protocol is designed to attempt to improve the current results of matched unrelated donor (MUD) allo bone marrow transplant (BMT) and will be a major step towards the introduction and refinement of graft engineering. Our approach will address in a rational fashion all major technical and clinical aspects of MUD allo BMT.
  Peripheral blood lymphocyte therapy; cyclophosphamide, tacrolimus, peripheral blood stem cell transplantation; total-body irradiation; 'allogeneic hematopoietic stem cell transplantation'
  Interventions: Procedure: peripheral blood lymphocyte therapy; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: total-body irradiation (TBI)

INTERVENTIONS:
Procedure: peripheral blood lymphocyte therapy — T-cell depletion will be accomplished using CD34 selection with the Baxter Isolex 300i v. 2.5 device. The desirable T-cell dose will be >0.5 x 105 but <1.0 x 105 CD3+ cells per kg. The targeted CD34 cell dose will be >2 x 106 cells/kg.
  Other Names: T-cell depletion
Procedure: allogeneic hematopoietic stem cell transplantation — Allogeneic Hematopoietic Stem Cell Transplantation
Procedure: peripheral blood stem cell transplantation — Peripheral blood stem cell transplantation
Radiation: total-body irradiation (TBI) — Treatment will be delivered using 6MV photons twice daily for 3 days

SUMMARY:
RATIONALE: Giving chemotherapy and total-body irradiation before a donor peripheral blood stem cell transplant helps stop the growth of cancer and abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. When stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Removing the T cells from the donor cells before transplant may stop this from happening. Giving an infusion of the donor's T cells (donor lymphocyte infusion) after the transplant may help destroy any remaining cancer cells (graft-versus-tumor effect).

PURPOSE: This phase II trial is studying T-cell depletion in donor stem cell transplant followed by delayed T cell infusions in treating patients with hematologic cancer or other disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine if T-cell depletion of a peripheral blood progenitor cell (PBPC) graft followed by delayed add-backs of defined doses of donor lymphocytes decreases the rate of graft-versus-host disease and its complications in matched unrelated donor (MUD) allogeneic peripheral blood progenitor cell (PBPC) transplantation in patients with hematologic cancers or other diseases.
* Determine whether targeted T-cell dosages in the PBPC graft can be achieved in these patients by positive CD34+ selection using the Baxter Inc. Isolex 300i v. 2.5.
* Determine the effects of T-cell depletion on the rate of engraftment in these patients.
* Develop a matched unrelated donor (MUD) allogeneic transplantation regimen that will decrease overall treatment-related mortality in these patients.

OUTLINE: This is a non-randomized study.

* Myeloablative preparative regimen: Patients receive cyclophosphamide IV once daily on days -5 and -4 followed by total body irradiation twice daily on days -3, -2, and -1. Patients also receive tacrolimus on day -1 administered by continuous IV infusion over 24 hours.
* Peripheral blood progenitor cell graft transplantation: Patients receive T-cell depleted, peripheral blood progenitor cells (PBPC) by IV infusion on day 0. Beginning 1 day after completion of the PBPC infusion, patients receive filgrastim (G-CSF) subcutaneously once daily until blood counts recover.
* Post transplantation T cell add-backs: Patients receive defined doses of donor T cells by IV infusion on days 45 and 100, in the absence of active graft-versus-host disease (GVHD) requiring steroids*.

NOTE: *A T cell add-back may be given in the presence of GVHD, if the investigator considers the risk from relapse or overwhelming viral infection to outweigh the risk of exacerbating GVHD.

Patients will be followed periodically for relapse and survival.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of any of the following hematologic cancers or other diseases:

  * Acute myelogenous leukemia

    * Relapsed or refractory disease with poor-risk cytogenetics
  * Acute lymphoblastic leukemia

    * Relapsed or refractory disease with poor-risk cytogenetics
  * Chronic myelogenous leukemia

    * Persistent disease after at least 6 months of treatment with imatinib mesylate (Gleevec)
  * Myelodysplasia, meeting 1 of the following criteria:

    * French-American-British Classification of refractory anemia with excess blasts (RAEB) or RAEB with transformation
    * International Prognostic Scoring System score > 2
  * Lymphoid malignancies, including non-Hodgkin lymphoma, Hodgkin disease, chronic lymphocytic leukemia, and prolymphocytic leukemia

    * Relapsed or refractory disease after at least 1 prior therapy
  * Myelofibrosis

    * Transfusion dependent (RBC's, platelets, or both)
  * Paroxysmal nocturnal hemoglobinuria (transfusion dependent)
  * Myeloproliferative disorder
  * Eosinophilic leukemia
  * Severe aplastic anemia

    * Corrected reticulocyte count < 1%
    * Platelet count < 30,000/mm³ (untransfused)
    * Bone marrow biopsy with < 15% cellularity
  * Plasma cell leukemia
* No essential thrombocytopenia or polycythemia vera
* No matched related donor available
* Must have an 8/8 or 7/8 serologic HLA matched unrelated donor available

PATIENT CHARACTERISTICS:

* Cardiac ejection fraction ≥ 45% (if < 45%, then cardiac consult required)
* Not pregnant or nursing
* Negative pregnancy test
* FEV_1 and DLCO ≥ 45% predicted
* Creatinine < 2.0 mg/dL
* Bilirubin < 2.0 mg/dL
* HIV negative

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior allogeneic bone marrow transplantation
* No concurrent administration of steroids with T-cell add-backs

INCLUSION CRITERIA:

* Patient actual weight must not be greater than 1.5x their ideal body weight
* Cardiac ejection fraction >45%. If less than 45%, a Cardiac consult will be obtained.
* A suitably matched unrelated donor that is at least a 7 out of 8 HLA serologic match.
* Patient is not pregnant.
* FEV 1 and DLCO > 45% predicted on pulmonary function testing.
* Serum creatinine <2.0 mg/dl, serum bilirubin <2.0 mg/dl.
* Patient and donor are HIV negative.
* Diagnosis of one of the following diseases
* Acute myelogenous leukemia
* Relapsed disease,
* Refractory disease, or
* With poor-risk cytogenetics
* Acute lymphoblastic leukemia
* Relapsed disease,
* Refractory disease, or
* With poor-risk cytogenetics
* Chronic myelogenous leukemia
* Persistent disease after at least 6 months of treatment with Imatinib Mesylate (Gleevec)
* Myelodysplasia
* FAB Classification of RAEB or RAEB-T -Or-
* IPSS score >2
* Lymphoid malignancies, including non-Hodgkin's lymphoma, Hodgkin's disease, chronic lymphocytic leukemia and prolymphocytic leukemia
* Relapsed or refractory disease after at least 1 prior therapy
* Myelofibrosis
* Transfusion dependence (RBC's, platelets, or both)
* Paroxysmal Nocturnal Hemoglobinuria (PNH)
* Transfusion dependent
* Myeloproliferative Disorder
* Eosinophilic Leukemia
* Severe aplastic anemia (<1% corrected reticulocyte count, <30,000 untransfused platelet count, bone marrow biopsy with <15% cellularity)
* Plasma cell leukemia
* Patients with ET or PV will not be candidates unless their disease has transformed to end stage myelofibrosis or acute leukemia, for which eligibility criteria for myelofibrosis or acute leukemia would apply.
* Patient must signed written informed consent.

EXCLUSION CRITERIA:

* Inability to give informed consent
* Absence of any of the above mentioned medical conditions
* Availability of matched-related donor
* History of prior allogeneic BMT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2004-01; Primary Completion 2009-08 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian J. Bolwell, MD, Study Chair — The Cleveland Clinic; Jarek Maciejewski, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from local hospital from January, 2006 through January, 2009.
Groups:
- T-Cell Depletion Transplant: Our protocol is designed to attempt to improve the current results of MUD allo BMT and will be a major step towards the introduction and refinement of graft engineering. Our approach will address in a rational fashion all major technical and clinical aspects of MUD allo BMT.
  Peripheral blood lymphocyte therapy; cyclophosphamide, tacrolimus, peripheral blood stem cell transplantation; total-body irradiation; 'allogeneic hematopoietic stem cell transplantation'
  peripheral blood lymphocyte therapy: T-cell depletion
  cyclophosphamide: T-cell depletion
  tacrolimus: T-cell depletion
  allogeneic hematopoietic stem cell transplantation: T-cell depletion
  peripheral blood stem cell transplantation: T-cell depletion
  total-body irradiation: T-cell depletion
Period: Overall Study
Arm/Group | T-Cell Depletion Transplant
Started | 13
Completed | 12
Not Completed | 1
Not completed — Did not collect enough CD34+ cells | 1

BASELINE CHARACTERISTICS:
Arm/Group | T-Cell Depletion Transplant
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 46 [18 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Treatment-related Mortality (TRM)
Description: The complication rate in matched unrelated donor (MUD) allogeneic bone marrow transplant (allo BMT) is known to be high. Graft failure and severe graft versus host disease (GvHD) are the most significant contributors to treatment related mortality (TRM). This treatment regimen will be considered unacceptable if the number of patients that experience TRM is 55% or greater, and effective if TRM is 33% or less.
Time Frame: 180 days after transplant
Population: Patients that received treatment
Measure: Number; unit: participants
Arm/Group | T-Cell Depletion Transplant
Number analyzed (Participants) | 12
participants | 8

2. Secondary Outcome: The Rate of Acute Graft Versus Host Disease (GVHD)
Time Frame: D+100 from transplant
Measure: Number; unit: participants
Groups:
- T-Cell Depletion Transplant: Our protocol is designed to attempt to improve the current results of matched unrelated donor allogeneic bone marrow transplant (MUD allo BMT) and will be a major step towards the introduction and refinement of graft engineering. Our approach will address in a rational fashion all major technical and clinical aspects of MUD allo BMT.
  Peripheral blood lymphocyte therapy; cyclophosphamide, tacrolimus, peripheral blood stem cell transplantation; total-body irradiation; allogeneic hematopoietic stem cell transplantation;
  peripheral blood lymphocyte therapy: T-cell depletion
  cyclophosphamide: T-cell depletion
  tacrolimus: T-cell depletion
  allogeneic hematopoietic stem cell transplantation: T-cell depletion
  peripheral blood stem cell transplantation: T-cell depletion
  total-body irradiation: T-cell depletion
Arm/Group | T-Cell Depletion Transplant
Number analyzed (Participants) | 12
participants | 11

3. Secondary Outcome: Number of Participants With Duration of Absolute Neutropenia
Time Frame: D+100 from transplant
Measure: Number; unit: participants
Groups:
- T-Cell Depletion Transplant: peripheral blood lymphocyte therapy: T-cell depletion will be accomplished using CD34 selection with the Baxter Isolex 300i v. 2.5 device. The desirable T-cell dose will be >0.5 x 105 but <1.0 x 105 CD3+ cells per kg. The targeted CD34 cell dose will be >2 x 106 cells/kg.
  cyclophosphamide: Cyclophosphamide 60 mg/kg/d for 2 days on Day -5 and Day -4
  tacrolimus: tacrolimus on day -1 administered by continuous IV infusion over 24 hours
  allogeneic hematopoietic stem cell transplantation
  peripheral blood stem cell transplantation
  total-body irradiation (TBI): Treatment will be delivered using 6MV photons twice daily for 3 days
Arm/Group | T-Cell Depletion Transplant
Number analyzed (Participants) | 12
participants | 10

4. Secondary Outcome: Number of Participants Able to Receive T-cell Add Backs
Description: Patients receive defined doses of donor T cells by IV infusion on days 45 and 100, in absence of active graft-versus-host disease (GVHD) requiring steroids.
Time Frame: through D+100
Measure: Number; unit: participants
Arm/Group | T-Cell Depletion Transplant
Number analyzed (Participants) | 12
participants | 3

5. Secondary Outcome: Number of Participants With Relapse-free Survival
Description: number of patients that were still alive and relapse free
Time Frame: after 7 years of follow up
Population: All patients that received treatment
Measure: Number; unit: participants
Arm/Group | T-Cell Depletion Transplant
Number analyzed (Participants) | 12
participants | 2

ADVERSE EVENTS:
Time Frame: Adverse events data was over the course of the study for approximately 7 years
Groups:
- T-Cell Depletion Transplant: peripheral blood lymphocyte therapy: T-cell depletion
  cyclophosphamide: T-cell depletion
  tacrolimus: T-cell depletion
  allogeneic hematopoietic stem cell transplantation: T-cell depletion
  peripheral blood stem cell transplantation: T-cell depletion
  total-body irradiation: T-cell depletion
Arm/Group | T-Cell Depletion Transplant
Serious Adverse Events (participants affected / at risk) | 9/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-Cell Depletion Transplant (N=12)
Death by Relapse (General disorders) | 4 (4)
Death from Acute GVHD (General disorders) | 3 (3)
Death due to respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death due to Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-Cell Depletion Transplant (N=12)
Hospitalization for fever (General disorders) | 7 (24)
Hospitalized with hypoglycemia (Endocrine disorders) | 1 (1)
Hospitalized with GVHD (General disorders) | 7 (11)
Hospitalized with mental status changes (Nervous system disorders) | 2 (2)
Hospitalized with Infection (Infections and infestations) | 9 (38)
Hospitalized for Nausae, Vomiting and Diarrhea (General disorders) | 5 (22)
Hospitalized for respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalized for broken leg (General disorders) | 1 (1)
Hospitalized for shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalized for hypertension (General disorders) | 1 (1)
Hospitalized for chest pains (Cardiac disorders) | 1 (1)
Hospitalized for Syncope and dizziness (General disorders) | 1 (1)
Hospitalized for abdominal pain (Gastrointestinal disorders) | 2 (4)
Hospitalized for puritus and plolyarthagias (General disorders) | 1 (1)
Hospitalized for pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalized for abscess (Infections and infestations) | 2 (2)
Hospitalized for blood in stool and (Gastrointestinal disorders) | 1 (2)
Hospitalized for TTP (Thrombotic Thrombocytopenic Purpura) (Blood and lymphatic system disorders) | 1 (1)
Hospitalized for muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2)
Hospitalized for relapse of disease (General disorders) | 1 (1)
Hospitalized for a motor vehicle accident (Injury, poisoning and procedural complications) | 1 (1)
Hospitalized for necrosis of knees (Musculoskeletal and connective tissue disorders) | 1 (1)
Hospitalized for knee replacement (Surgical and medical procedures) | 1 (2)
Hospitalized for numbness in hands and feet (General disorders) | 1 (1)
Hospitalized for surgery medial epicondylitis (Surgical and medical procedures) | 1 (1)
Hospitalized for mucocitus and rash (Skin and subcutaneous tissue disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Hospitalized for dysuria (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No